CLINICAL TRIAL: NCT05529849
Title: A Two-Part Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Subcutaneous Doses of TCMCB07 on Healthy Male and Female Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of TCMCB07 in Single and Multiple Ascending Doses in Health Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endevica Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 205823
Record Dates: First submitted 2022-07-28; First posted 2022-09-07 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TCMCB07 (Experimental): once daily subcutaneous injection
  Interventions: Drug: TCMCB07
- Placebo (Placebo Comparator): once daily subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TCMCB07 — Subcutaneous injection of TCMCB07
  Arms: TCMCB07
Drug: Placebo — Matching subcutaneous placebo
  Arms: Placebo

SUMMARY:
This study will test an experimental drug named TCMCB07 for the treatment of cancer cachexia. Cachexia is a syndrome characterized by weight loss, anorexia, weakness or lack of energy, and anemia. Cachexia occurs in many cancers, usually at the advanced stages of disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females (WONCBP), aged 18 to 55 years inclusive, at time of signing informed consent.
* Body mass index 18.0 to 30.0 kg/m2 as measured at Screening or, if outside this range, considered not clinically significant by the investigator.
* Weight ≥ 50 kg at Screening

Exclusion Criteria:

* Serious adverse reaction or serious known hypersensitivity to melanocortins or polyethylene glycol.
* Evidence of current severe acute respiratory syndrome coronavirus 2 infection.
* Clinically significant abnormal clinical chemistry, hematology, or urinalysis as judged by the investigator.
* Subjects who have received any IP in a clinical research study within 5 half-lives or within 30 days prior to first dose. However, in no event shall the time between last receipt of IP and first dose be less than 30 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Number of people with an Adverse Event Assessment | 6 Months
  Adverse Event monitoring
Number of participants with abnormal vital signs | 6 Months
  Assessment of vital signs
Number of people with abnormal laboratory test results | 6 Months
  Analysis of clinical chemistry, hematology, and urinalysis
Number of people with abnormal Electrocardiograms | 6 Months
  12-lead ECGs will be used and an assessment of any clinically significant abnormality from baseline will be reported as an AE
Number of people with abnormal physical examinations | 6 Months
  Physical and injection site examination

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 6 Months
  Non-compartmental techniques will be employed to obtain estimates of cmax
Area under the plasma concentration versus time curve (AUC) | 6 months
  Non-compartmental techniques will be employed to obtain estimates of AUC

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bermudez, MD, CPI, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences -- Miami, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.endevicabio.com